CLINICAL TRIAL: NCT06491134
Title: Phase Ib Trial of Liposomal Irinotecan With Cisplatin and Concurrent Radiotherapy in Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Liposomal Irinotecan With Cisplatin and Concurrent Radiotherapy in Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Jun wang, offices director, Hebei Medical University Fourth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HESS-LAEC-202401
Record Dates: First submitted 2024-06-27; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: liposomal irinotecan; Cisplatin; Radiotherapy; Locally Advanced Esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- liposomal irinotecan (Experimental): liposomal irinotecan With Cisplatin and Concurrent Radiotherapy
  Interventions: Drug: Liposomal Irinotecan Hydrochloride

INTERVENTIONS:
Drug: Liposomal Irinotecan Hydrochloride — liposomal irinotecan With Cisplatin and Concurrent Radiotherapy

SUMMARY:
Observation of maximum tolerable dose (MTD), dose limiting toxicity (DLT), and phase II clinical recommended dose (RP2D) of liposomal irinotecan With Cisplatin and Concurrent Radiotherapy in Locally Advanced Esophageal squamous cell carcinoma. Evaluate the efficacy and safety of liposomal irinotecan With Cisplatin and Concurrent Radiotherapy in the treatment of locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and be willing to sign written informed consent and be able to follow research protocols for treatment.
2. Age 18-75 years.
3. Histologically confirmed cT2-T4a,N0-N+,M0 Esophageal Squamous Carcinoma.
4. Existence of measurable and/or unmeasurable lesions that meet the criteria for evaluating the efficacy of solid tumors (RECIST 1.1)
5. No previous anti-tumor therapy for esophageal cancer
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
7. Life expectancy ≥ 3months
8. Adequate organ and bone marrow function measured within14 days prior to administration of study treatment as defined below:

   Haemoglobin ≥ 90g/dL Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L Total bilirubin ≤institutional upper limit of normal Aspartate aminotransferase (AST(SGOT)/Alanine transaminase (ALT)SGPT) ≤ 2.5 x institutional upper limit of normal Serum creatinine ≤ 1.2mg/dL And creatinine clearance ≥50mL/min (Cockcroft-Gault formula)
9. Women who are not pregnant or lactating. During the study period and within 6 months of the end of the study treatment, childbearing age Women/men should take effective contraceptive measures.

Exclusion Criteria:

1. patients with other malignant tumors within the previous 5 years, except for cure carcinoma in situ, skin basal cell carcinoma.
2. Allergic to cisplatin.
3. Patients with a history of esophageal squamous cell carcinoma surgery.
4. A history of fistula caused by primary tumor infiltration.
5. Have higher, esophageal fistula or esophageal perforation of gastrointestinal bleeding risk.
6. Poor nutritional status, BMI < 18.5kg/m2, or PG-SGA score ≥9.
7. Pulmonary fibrosis or interstitial pneumonia was diagnosed within 28 days before enrollment.
8. Patients with active hepatitis B, hepatitis C, syphilis.
9. major cardiovascular disease, including any of the following:

   1. Within 6 months before enrollment, congestive heart failure (defined as New York Heart Association grade III or IV), myocardial infarction, unstable angina, coronary angioplasty, stenting, coronary artery bypass grafting, cerebrovascular accident, or hypertensive crisis.
   2. A history of clinically significant ventricular arrhythmias
   3. Friderica-modified QT interval >450 msec in men and >470 msec in women
   4. History of congenital long QT syndrome or family history
   5. Arrhythmias requiring antiarrhythmic drug therapy
   6. History of deep vein thrombosis, pulmonary embolism, or any other major thromboembolism within 3 months before enrollment
10. Severe prolonged diarrhoea.
11. Severe mental illness.
12. Use of strong inhibitors or inducers such as CYP3A4, CYP2C8 and UGT1A1.
13. Participate in other trials within 4 weeks before the start of the trial.
14. The investigators believe that patients were inappropriate for participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-06-27 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
maximum tolerable dose (MTD) | through study completion, an average of 1 year
  The maximum tolerated dose/maximum administered dose will be determined by the number of participants experiencing dose-limiting

SECONDARY OUTCOMES:
Objective response rate (ORR) | Within 28 days of the end of treatment
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR
Progress-free survival(PFS) | 2-years
  Progression-free survival will be measured from the start of treatment until the first documentation of confirmed disease progression or death due to any cause, whichever occurs first.

IPD SHARING:
Plan to Share IPD: No